CLINICAL TRIAL: NCT02009332
Title: A Combined Phase 1 and Phase 2 Study of Albumin-bound Rapamycin Nanoparticles (Nab-rapamycin, ABI-009) in the Treatment of BCG Refractory or Recurrent Nonmuscle Invasive Transitional Cell Bladder Cancer
Brief Title: Phase 1/2 Study of ABI-009 in Nonmuscle Invasive Bladder Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Aadi Bioscience, Inc. (Industry)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: BC001; 1R42CA171552-01 (NIH)
Record Dates: First submitted 2013-12-08; First posted 2013-12-12 (Estimated); Results first posted 2021-06-08 (Actual); Last update posted 2021-06-08 (Actual); Status verified 2021-05

CONDITIONS: Non-muscle Invasive Bladder Cancer (NMIBC)
MeSH Terms: conditions — Non-Muscle Invasive Bladder Neoplasms | interventions — Gemcitabine

STUDY DESIGN:
Intervention Model Description: The phase 1 dose-escalation portion used the 3+3 dose escalation rule. Initially 3 patients will be treated. If none develops DLT following the third weekly instillation, the dose can be escalated. If only 1 of the first 3 patients develops DLT, then an additional 3 patients will be treated at that dose. At any dose level, if 2 or more cases develop DLT, the prior dose will be defined as the MDD once 6 patients have been treated at this level with less than 2 patients experiencing a DLT.
  In phase 2, up to 29 patients will receive intravesical ABI-009 and gemcitabine using the Simon 2-stage design: initially, there will be only 10 patients enrolled with a rejection rule that only if there are 2 or more positive responses will the study proceed to further enrollment of the next 19 patients.
Oversight: Data Monitoring Committee: Yes

ARMS (6):
- Phase 1: ABI-009 100 mg/week (Experimental): Phase 1, Cohort 1: ABI-009 injectable suspension, 100 mg in 80 mL 0.9% saline, administered intravesically and retained for 2 hours, once per week for 6 weeks
  Interventions: Drug: ABI-009
- Phase 1: ABI-009 200 mg/week (Experimental): Phase 1, Cohort 2: ABI-009 injectable suspension, 200 mg in 80 mL 0.9% saline, administered intravesically and retained for 2 hours, once per week for 6 weeks
  Interventions: Drug: ABI-009
- Phase 1: ABI-009 100 mg 2×/week (Experimental): Phase 1, Cohort 2b: ABI-009 injectable suspension, 100 mg in 80 mL 0.9% saline, administered intravesically and retained for 2 hours, twice per week (total dose 200 mg per week) for 6 weeks
  Interventions: Drug: ABI-009
- Phase 1: ABI-009 300 mg/week (Experimental): Phase 1, Cohort 3: ABI-009 injectable suspension, 300 mg in 80 mL 0.9% saline, administered intravesically and retained for 2 hours, once per week for 6 weeks
  Interventions: Drug: ABI-009
- Phase 1: ABI-009 400 mg/week (Experimental): Phase 1, Cohort 4: ABI-009 injectable suspension, 400 mg in 80 mL 0.9% saline, administered intravesically and retained for 2 hours, once per week for 6 weeks
  Interventions: Drug: ABI-009
- Phase 2: ABI-009 400 mg/week + Gemcitabine 2000 mg/week (Experimental): ABI-009 injectable suspension, 200 mg in 80 mL 0.9% saline, administered intravesically and retained for 1 hour, once per week for 6 weeks; Gemcitabine, 2000 mg in 100 mL saline, administered intravesically after voiding of ABI-009 and retained for 1 hour, once per week for 6 weeks
  Interventions: Drug: ABI-009; Drug: Gemcitabine

INTERVENTIONS:
Drug: ABI-009 — ABI-009 is a nanoparticle albumin-bound (nab®) formulation of the mammalian Target of Rapamycin ( mTOR) inhibitor, sirolimus. Specifically, ABI-009 is a sterile lyophilized powder of albumin-bound sirolimus nanoparticles with a mean particle size of less than 100 nm.
  Other Names: nab-sirolimus; nab-rapamycin
Drug: Gemcitabine — Gemcitabine is administered after ABI-009 in the Phase 2 study.
  Arms: Phase 2: ABI-009 400 mg/week + Gemcitabine 2000 mg/week

SUMMARY:
Purpose of this study is to determine appropriate dosing of ABI-009 and evaluate the safety and anti-tumor activity of ABI-009 in treatment of non-muscle invasive bladder cancer

ELIGIBILITY:
Inclusion Criteria:

1. Patients must have a diagnosis of transitional cell carcinoma (TCC) of the urinary bladder confirmed at the study institution. The patient must have demonstrated nonmuscle-invasive bladder cancer refractory or recurrent to standard intravesical therapy. Refractory disease is defined as failure to achieve tumor-free status by 6 months of initiation of adequate BCG therapy. Recurrent disease is defined as reappearance of disease after achieving a tumor-free status by 6 months of initiation of adequate BCG therapy. Adequate BCG therapy includes at least 6 weeks induction plus 3 additional doses of either induction or maintenance. Patients with a history of other intravesical agents (except nab-rapamycin or gemcitabine) in addition to standard BCG will also be allowed to enroll. All grossly visible disease must be fully resected and pathologic stage will be confirmed at the institution where the patient is enrolled. This will include stage Ta, T1, Tis and exclude all patients with muscle invasion (T2).

   1. For phase 1, patients with multifocal low-grade Ta histology will be eligible for participation
   2. For phase 2, individuals with Ta disease only must have documentation of high-grade histology
   3. For phase 2, prior intravesical treatment with nab-rapamycin or gemcitabine is not allowed
2. Age >18 and must be able to read, understand, and sign informed consent
3. Performance Status: ECOG 0, 1, and 2 (See Appendix III)
4. Hematologic inclusion within 2 weeks of start of treatment

   1. Absolute neutrophil count >1,500/mm3
   2. Hemoglobin >9.0 g/dl
   3. Platelet count >100,000/mm3
5. Hepatic inclusion within 2 weeks of entry

   1. Total bilirubin must be within normal limits.
   2. Adequate renal function with serum creatinine ≤2.5 mg/dL
   3. Aspartate transaminase (AST) and alanine transaminase (ALT) ≤2.5 x ULN for the institution, alkaline phosphatase ≤ 2.5 x ULN for the institution, unless bone metastasis is present in the absence of liver metastasis
6. Women of childbearing potential must have a negative pregnancy test.
7. All patients of childbearing potential must be willing to consent to using effective contraception, ie, intrauterine device, birth control pills, depo-provera, and condoms while on treatment and for 3 months after their participation in the study ends.

Exclusion Criteria:

1. Any other malignancy diagnosed within 1 year of study entry (except basal or squamous cell skin cancers or noninvasive cancer of the cervix) is excluded
2. Concurrent treatment with any chemotherapeutic agent
3. Women who are pregnant or lactating
4. History of vesicoureteral reflux or an indwelling urinary stent
5. Participation in any other research protocol involving administration of an investigational agent within 1 month prior to study entry
6. History of radiation to the pelvis
7. History of interstitial lung disease and/or pneumonitis
8. Evidence of metastatic disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2014-04-09 (Actual); Primary Completion 2019-12-01 (Actual); Study Completion 2019-12-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James McKiernan, MD, Principal Investigator — Columbia University
Locations (2):
- United States (2):
  - Columbia University Medical Center, New York, New York
  - Vanderbilt University Medical Center, Nashville, Tennessee

RESULTS

PARTICIPANT FLOW:
Groups:
- Phase 2: ABI-009 200 mg/Week + Gemcitabine 2000 mg/Week: ABI-009 injectable suspension, 200 mg in 80 mL 0.9% saline, administered intravesically and retained for 1 hour, once per week for 6 weeks; Gemcitabine, 2000 mg in 100 mL saline, administered intravesically after voiding of ABI-009 and retained for 1 hour, once per week for 6 weeks
Period: Phase 1: Dose Level 1 (Weeks 1-10)
Arm/Group | Phase 1: ABI-009 100 mg/Week | Phase 1: ABI-009 200 mg/Week | Phase 1: ABI-009 100 mg 2×/Week | Phase 1: ABI-009 300 mg/Week | Phase 1: ABI-009 400 mg/Week | Phase 2: ABI-009 200 mg/Week + Gemcitabine 2000 mg/Week
Started | 3 | 0 | 0 | 0 | 0 | 0
Completed | 3 (Cohort 1 completed 6-week treatment.) | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Phase 1: Dose Level 2/2b (Wks 11-29)
Arm/Group | Phase 1: ABI-009 100 mg/Week | Phase 1: ABI-009 200 mg/Week | Phase 1: ABI-009 100 mg 2×/Week | Phase 1: ABI-009 300 mg/Week | Phase 1: ABI-009 400 mg/Week | Phase 2: ABI-009 200 mg/Week + Gemcitabine 2000 mg/Week
Started | 0 | 4 | 1 | 0 | 0 | 0
Completed | 0 | 3 (Cohort 2 completed 6-week treatment.) | 1 (Cohort 2b stopped due to lack of enrollment.) | 0 | 0 | 0
Not Completed | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Physician Decision | 0 | 1 | 0 | 0 | 0 | 0
Period: Phase 1: Dose Level 3 (Weeks 30-47)
Arm/Group | Phase 1: ABI-009 100 mg/Week | Phase 1: ABI-009 200 mg/Week | Phase 1: ABI-009 100 mg 2×/Week | Phase 1: ABI-009 300 mg/Week | Phase 1: ABI-009 400 mg/Week | Phase 2: ABI-009 200 mg/Week + Gemcitabine 2000 mg/Week
Started | 0 | 0 | 0 | 3 | 0 | 0
Completed | 0 | 0 | 0 | 3 (Cohort 3 completed 6-week treatment.) | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Phase 1: Dose Level 4 (Weeks 48-77)
Arm/Group | Phase 1: ABI-009 100 mg/Week | Phase 1: ABI-009 200 mg/Week | Phase 1: ABI-009 100 mg 2×/Week | Phase 1: ABI-009 300 mg/Week | Phase 1: ABI-009 400 mg/Week | Phase 2: ABI-009 200 mg/Week + Gemcitabine 2000 mg/Week
Started | 0 | 0 | 0 | 0 | 4 | 0
Completed | 0 | 0 | 0 | 0 | 3 (Cohort 4 completed 6-week treatment.) | 0
Not Completed | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 1 | 0
Period: Phase 2 (Weeks 206-252)
Arm/Group | Phase 1: ABI-009 100 mg/Week | Phase 1: ABI-009 200 mg/Week | Phase 1: ABI-009 100 mg 2×/Week | Phase 1: ABI-009 300 mg/Week | Phase 1: ABI-009 400 mg/Week | Phase 2: ABI-009 200 mg/Week + Gemcitabine 2000 mg/Week
Started | 0 | 0 | 0 | 0 | 0 | 6
Completed | 0 | 0 | 0 | 0 | 0 | 5 (Phase 2 stopped due to lack of efficacy.)
Not Completed | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Phase 1: ABI-009 100 mg 2x/Week: Phase 1, Cohort 2b: ABI-009 injectable suspension, 100 mg in 80 mL 0.9% saline, administered intravesically and retained for 2 hours, twice per week (total dose 200 mg per week) for 6 weeks
- Phase 2, Efficacy: ABI-009 injectable suspension, 200 mg in 80 mL 0.9% saline, administered intravesically and retained for 1 hour, once per week for 6 weeks; Gemcitabine, 2000 mg in 100 mL saline, administered intravesically after voiding of ABI-009 and retained for 1 hour, once per week for 6 weeks
- Total: Total of all reporting groups
Arm/Group | Phase 1: ABI-009 100 mg/Week | Phase 1: ABI-009 200 mg/Week | Phase 1: ABI-009 100 mg 2x/Week | Phase 1: ABI-009 300 mg/Week | Phase 1: ABI-009 400 mg/Week | Phase 2, Efficacy | Total
Number analyzed (Participants) | 3 | 4 | 1 | 3 | 4 | 6 | 21
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 0 | 3 | 0 | 0 | 0 | 0 | 3
  >=65 years | 3 | 1 | 1 | 3 | 4 | 6 | 18
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 0 | 0 | 0 | 0 | 1 | 2
  Male | 2 | 4 | 1 | 3 | 4 | 5 | 19
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0 | 0 | 0
  White | 3 | 4 | 1 | 3 | 4 | 6 | 21
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 3 | 4 | 1 | 3 | 4 | 6 | 21

OUTCOME MEASURES:

1. Primary Outcome: Phase 1: Dose Limiting Toxicities (DLT) Following Intravesical Administration of ABI-009
Description: The primary endpoint of the Phase 1 study is DLT following intravesical administration of ABI-009 in patients with BCG refractory or recurrent nonmuscle-invasive transitional cell carcinoma (TCC) of the bladder to identify maximum deliverable dose (MDD). Systemic DLT will be defined as any grade systemic toxicity using the NCI CTCAE version 4.0. Local dose limiting toxicity was defined as grade 3 or 4 bladder toxicity (hematuria, dysuria, urinary retention, urinary frequency/urgency, or bladder spasms) using the NCI CTCAE version 4.0.
Time Frame: Duration of treatment (6 weeks) plus 30 days follow up (up to 2.5 months)
Population: All Phase 1 patients who received at least 1 treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 1: ABI-009 100 mg/Week | Phase 1: ABI-009 200 mg/Week | Phase 1: ABI-009 100 mg 2×/Week | Phase 1: ABI-009 300 mg/Week | Phase 1: ABI-009 400 mg/Week
Number analyzed (Participants) | 3 | 4 | 1 | 3 | 4
Participants | 0 | 0 | 0 | 0 | 0
Statistical Analysis 1: Comparison: Phase 1: ABI-009 100 mg/Week vs Phase 1: ABI-009 200 mg/Week vs Phase 1: ABI-009 100 mg 2×/Week vs Phase 1: ABI-009 300 mg/Week vs Phase 1: ABI-009 400 mg/Week; Test type: Other; maximum deliverable dose (MDD) = 400 — Maximum deliverable dose (MDD) was not reached in the Phase 1 study as no DLTs were observed in any of the dose groups up to ABI-009 400 mg/week

2. Primary Outcome: Phase 2: Number of Participants Achieving a Complete Response Following Intravesical Administration of ABI-009 and Gemcitabine
Description: The primary objective of the Phase 2 study is to evaluate the utility (potential for clinical efficacy) of ABI-009 in combination with gemcitabine in the treatment of BCG refractory or recurrent nonmuscle-invasive TCC of the bladder. Response rate will be measured and documented at the 6-week post-treatment assessment, including cystoscopy with biopsy. A complete response is defined as a cancer-negative biopsy at the 6-week post-treatment cystoscopy. No response will be defined as positive cystoscopic biopsy.
Time Frame: End of Study [EOS, 3 months]
Population: Analysis population includes all patients who have completed the planned 6 treatment cycles and have 6 week follow up cystoscopy data available
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 2: ABI-009 400 mg/Week + Gemcitabine 2000 mg/Week
Number analyzed (Participants) | 5
Participants | 1

3. Secondary Outcome: Phase 1: Number of Participants Achieving a Complete Response Following Intravesical Administration of ABI-009
Description: Response rate will be measured and documented at the 6-week post-treatment assessment, including cystoscopy with biopsy. A complete response is defined as a cancer-negative biopsy at the 6-week post-treatment cystoscopy. No response will be defined as positive cystoscopic biopsy.
Time Frame: End of Study [EOS, 3 months]
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 1: ABI-009 100 mg/Week | Phase 1: ABI-009 200 mg/Week | Phase 1: ABI-009 100 mg 2×/Week | Phase 1: ABI-009 300 mg/Week | Phase 1: ABI-009 400 mg/Week
Number analyzed (Participants) | 3 | 3 | 1 | 3 | 3
Participants | 0 | 1 | 0 | 0 | 1

ADVERSE EVENTS:
Time Frame: From the signing of the informed consent through the 6-week induction treatment period and the 30-day follow-up period (up to 2.5 months). An additional 4 months for patients who received 3 additional monthly maintenance treatments (up to 6.5 months).
Arm/Group | Phase 1: ABI-009 100 mg/Week | Phase 1: ABI-009 200 mg/Week | Phase 1: ABI-009 100 mg 2×/Week | Phase 1: ABI-009 300 mg/Week | Phase 1: ABI-009 400 mg/Week | Phase 2: ABI-009 400 mg/Week + Gemcitabine 2000 mg/Week
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/4 | 0/1 | 0/3 | 0/4 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/4 | 0/1 | 0/3 | 0/4 | 0/6
Other Adverse Events (participants affected / at risk) | 2/3 | 1/4 | 1/1 | 3/3 | 3/4 | 6/6
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase 1: ABI-009 100 mg/Week (N=3) | Phase 1: ABI-009 200 mg/Week (N=4) | Phase 1: ABI-009 100 mg 2×/Week (N=1) | Phase 1: ABI-009 300 mg/Week (N=3) | Phase 1: ABI-009 400 mg/Week (N=4) | Phase 2: ABI-009 400 mg/Week + Gemcitabine 2000 mg/Week (N=6)
Hematuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 0 (0)
Urinary tract infection (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 2 (2)
Penis Lesion/rash (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Increased frequency and urgency of urination (Renal and urinary disorders) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 1 (1)
Abnormal urine analysis (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Dysuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Incontinence (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Inguinal and thigh pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Kidney stone (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Prostatitis (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Anemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (2)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Decreased absolute neutrophil (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Decreased white blood cell (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Elevated bilirubin (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Elevated creatinine (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bladder spasm (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 5 (21)
Urinary tract pain (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (9)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Worsening of congestive heart failure (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Worsening of chronic kidney disease (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Worsening of edema of extremities (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Mucositis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3)
Upper respiratory tract infection (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Fever (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Malaise (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hyponatremia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-04-20): https://cdn.clinicaltrials.gov/large-docs/32/NCT02009332/Prot_SAP_000.pdf